CLINICAL TRIAL: NCT04764383
Title: Histaminergic Basis of Fatigue in Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn as more data drug analysis is recommended before the study.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kottil W. Rammohan, Professor of Clinical Neurology, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20201550
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Histamine
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Histidine; Histamine; Carbidopa

STUDY DESIGN:
Intervention Model Description: double-blind randomized cross-over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PK/PD Group (Experimental): Participants in the Pharmacokinetic (PK)/pharmacodynamic (PD) Group will receive L-Histidine and Lodosyn daily for 7 consecutive days.
  Interventions: Drug: L-Histidine; Drug: Lodosyn
- L-Histidine and Lodosyn followed by Placebo Group (Placebo Comparator): Participants in this group will receive L-Histidine and Lodosyn daily for 2 consecutive weeks followed by Placebo for an additional 2 consecutive weeks with a 1-week wash-out period in between.
  Interventions: Drug: L-Histidine; Drug: Placebo; Drug: Lodosyn
- Placebo followed by L-Histidine and Lodosyn Group (Experimental): Participants in this group will receive Placebo daily for 2 consecutive weeks followed by L-Histidine and Lodosyn for an additional 2 consecutive weeks with a 1 week wash out period in between.
  Interventions: Drug: L-Histidine; Drug: Placebo; Drug: Lodosyn

INTERVENTIONS:
Drug: L-Histidine — 1000 mg capsules taken by mouth (PO) twice daily (BID).
  Other Names: Histamine
Drug: Placebo — Microcrystalline cellulose (placebo) 1000 mg capsules taken by mouth (PO) twice daily (BID).
  Arms: L-Histidine and Lodosyn followed by Placebo Group; Placebo followed by L-Histidine and Lodosyn Group
Drug: Lodosyn — 50 mg capsules taken PO BID.

SUMMARY:
The purpose of this research study is to identify a way to improve the feeling of exhaustion that patients might experience because of Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion and Exclusion Criteria

For Healthy (Normal) Participants

Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60
* In good physical health without a history of chronic illness and considered generally healthy.

Exclusion Criteria:

* Adults unable to give informed consent due to cognitive impairment or mental disorders.
* Children below the age of consent
* Pregnant women (if the pregnancy test is positive during any stage of the study, subject will be removed from it)
* Prisoners
* Chronic untreated disorders like hypertension, diabetes, hyperlipidemia, depression, hypothyroidism etc., that could confound or interfere with the proposed therapy in the view of the PI are excluded. Stable treated above conditions are not exclusionary.
* Known chronic fatigue syndrome
* Blood disorders or coagulopathy
* Chronic allergies or history of asthma.
* Using antihistamines, bronchodilators or H2 blockers for hyperacidity
* Using medications for sleep, or known sleep disorders
* Any medication or condition deemed unsuitable by the PI. If necessary, subjects should wash out such medications for a duration of at least 5 half-lives.
* All medications prescribed and over the counter, should be approved by the PI during the duration of the trial.

For Multiple Sclerosis Participants

Inclusion Criteria:

* Established Multiple Sclerosis by McDonald Criteria - 2010 Revision or McDonald Criteria 2017. Relapsing-Remitting and progressive forms of MS are eligible
* Severe fatigue that has lasted greater than 6 months
* Clinically stable on a current therapy with any Disease Modifying Therapies (DMT)
* Fatigue Severity Score of >/= 4.0 will qualify as long as all other inclusion/exclusion criteria is met.

Exclusion Criteria:

* Adults unable to give informed consent due to cognitive impairment or mental disorders.
* Children below the age of consent
* Pregnant women (if the pregnancy test is positive during any stage of the study, subject will be removed from it)
* Prisoners
* Systemic disorders known to cause fatigue such as severe anemia, infections, chronic systemic infectious or inflammatory disorders, including known autoimmune disorders. (allowed as long is not present. Subject might qualify as per discretion of the Principal Investigator)
* Chronic fatigue syndrome
* Hypothyroidism (If treated and/or controlled subject might qualify as per discretion of the Principal Investigator)
* Systemic malignancy. Remote history of a malignancy is not a contraindication.
* Undergoing chemotherapy
* Depression (If treated and/or controlled subject might qualify as per discretion of the Principal Investigator)
* Sleep disorders including narcolepsy, excessive day-time sleep. (If treated and/or controlled subject might qualify as per discretion of the Principal Investigator)
* Ongoing substance abuse
* Excessive consumption of coffee or over-the-counter stimulants. Use of caffeine is not exclusionary but subjects are instructed to not change the use for the duration of the study.
* Concomitant medications of amantadine, methylphenidate, amphetamines, pemoline, barbiturates, tizanidine, MonoAmine Oxidase (MAO) inhibitors, benzodiazepines, barbiturates, tricyclic antidepressants, antihistamines, H2 blockers for Gastroesophageal reflux disease (GERD), Selective Serotonin Reuptake Inhibitor (SSRIs) and any other medication that in the opinion of the PI should be excluded. If used and approved by the PI at study entry, any change for the duration of the study is not permitted.
* Patients who were using modafinil for treatment of fatigues prior to the study may participate but will be required to undergo a washout of five half-lives prior to entry into the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 5 weeks
  Adverse events will be evaluated by treating physician.

SECONDARY OUTCOMES:
Efficacy as measured by FSS scores | Up to 5 weeks
  Efficacy will be reported as the number of participants that dropped one point or more from their baseline Fatigue Severity Scale (FSS) scores. FSS is a 9-item questionnaire with questions related to how fatigue interferes with certain activities according to a self-reported scale. Each of the items are scored on a 7 point scale with 1 = strongly disagree and 7 = strongly agree.
Efficacy as measured by MFIS Scores | Up to 5 weeks
  Modified Fatigue Impact Scale (MFIS) is a scale is used to measure fatigue with the total score ranging from 0 to 84 with 0 being the best possible score and 84 being the worst score.
Efficacy as measured by the VAS scores | Up to 5 weeks
  The Visual Analog Scale (VAS) allows participants to rate their health on a 20 cm vertical with a higher number indicating better outcomes.
Efficacy as measured by the MSQOL Scores | Up to 5 weeks
  Multiple Sclerosis Quality of Life (MSQOL) has a total score ranging from 0 to 100 with a higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kottil Rammohan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No